CLINICAL TRIAL: NCT04452526
Title: Improving Uptake of Cervical Cancer Prevention Services in Appalachia; Testing Multi-Level Interventions to Improve HPV Vaccination: The "I Vaccinate" Program
Brief Title: I Vaccinate: Testing Multi-Level Interventions to Improve HPV Vaccination
Acronym: IVaccinate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-20058; NCI-2020-01225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA229143 (NIH)
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cervical Carcinoma; Human Papillomavirus-Related Malignant Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM I (EARLY INTERVENTION) (educational material, reminders) (Experimental): Health systems receive educational materials consisting of posters, brochures and handouts. Providers complete survey about HPV knowledge, participate in educational session over 1 hour and receive educational handouts on the HPV vaccine. Patients receive educational materials about HPV vaccine and reminder letters for HPV vaccination
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Questionnaire Administration; Other: Reminder
- ARM II (DELAYED INTERVENTION)(education, reminder, usual care) (Experimental): Health systems, providers, and patients receive usual care for 12 months, then receive multi-level intervention as in Arm I.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Questionnaire Administration; Other: Reminder

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Other: Educational Intervention — Receive educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies
Other: Reminder — Receive reminder letter

SUMMARY:
This trial studies how well a multi-level health system-based intervention works in improving human papillomavirus (HPV) vaccine initiation and completion among children in health systems in four Appalachian states. Utilizing educational and promotional materials and electronic health record reminders, may improve the uptake of the HPV vaccine in children and young adults, ultimately preventing the development of cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Test the effectiveness of a multi-level intervention (MLI) directed at clinics, providers, and patients (parents of children aged 11-12) to improve HPV vaccine initiation and completion in health systems in four Appalachian states (Kentucky [KY], Ohio [OH], West Virginia [WV,] and Virginia [VA]) among children aged 11-12 and assess the effectiveness of the intervention program among subgroups, e.g., females versus (vs) males.

SECONDARY OBJECTIVES:

I. Assess sustainability of the intervention. II. Assess cost impacts of the intervention III. Assess changes in clinic practices that occur as a result of the intervention in terms of staff responsibilities for the vaccination process and reducing missed opportunities for vaccination.

IV. Assess whether interventions focused on 13-26 year olds increases catch-up vaccination.

V. Examine changes in knowledge and attitudes of providers via educational session pre-post surveys.

VI. Satisfaction with the intervention at the multiple levels.

OUTLINE: Health systems are randomized to 1 of 2 arms.

ARM I (EARLY INTERVENTION): Health systems receive educational materials consisting of posters, brochures and table tents. Providers complete survey about HPV knowledge, participate in educational session over 1 hour and receive educational handouts on the HPV vaccine. Patients receive educational materials about HPV vaccine and reminder letters for HPV vaccination.

ARM II (DELAYED INTERVENTION): Health systems, providers, and patients receive usual care for 12 months, then receive multi-level intervention as in Arm I.

ELIGIBILITY:
Inclusion Criteria:

CLINIC

* Located in one of the counties that are part of this program
* Provides care to patients aged 11-26
* Provides immunizations

HEALTH CARE PROVIDERS (PHYSICIANS, NURSES) AND OFFICE STAFF

* Practicing in a clinic in one of the participating health systems
* Personnel involved in the vaccine process (determined by individual clinics)
* Able to speak, read, and write English

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in rate of human papillomavirus (HPV) vaccination initiation among 11-12 year olds | Baseline up to 24 months
  The effectiveness of the intervention will be assessed by comparing early vs delayed intervention clinics at the end of the first implementation phase adjusting for baseline rates and pre- versus (vs) post implementation rates in the delayed implementation clinics.
Change in rate of HPV vaccination initiation among those 13-26 | Baseline up to 24 months
  The effectiveness of the intervention will be assessed by comparing early vs delayed intervention clinics at the end of the first implementation phase adjusting for baseline rates and pre- versus (vs) post implementation rates in the delayed implementation clinics.
Sustainability | Up to 24 months
  Will use logistic regression models with random health systems effects to compare odds of vaccination at the end of sustainability period to odds of vaccination at the end of the implementation period.
Cost-effectiveness | Up to 60 months
  Will conduct the cost-effectiveness analyses of using the multi-level intervention (MLI) intervention to promote HPV vaccination in three broad steps.
Change in knowledge of providers | Baseline up to 60 months
  Will compare changes in knowledge of providers via educational session pre-post survey. Changes in Knowledge following the educational session will be assessed using linear mixed models containing random health system effects.
Change in attitudes of providers | Baseline up to 60 months
  Will compare changes in attitudes of providers via educational session pre-post survey.

CONTACTS AND LOCATIONS:
Overall Officials: Electra D Paskett, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu